CLINICAL TRIAL: NCT06144853
Title: FDG-PET/CT as a Method of Patient Selection and Response Evaluation in Patients With Peritoneal Metastasis Treated With Pressurized IntraPeritoneal Aerosol Chemotherapy. A Pilot Study
Brief Title: The PIPAC-OPC7 Study: The Use of PET/CT Scans as a Method of Evaluation in Patients Treated With PIPAC, a Pilot Study.
Status: Recruiting | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PIPAC_OPC7
Record Dates: First submitted 2023-11-17; First posted 2023-11-22 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Peritoneal Cancer; Peritoneal Metastases; Peritoneal Carcinomatosis; Abdominal Cancer
Keywords: PIPAC; Pressurized intraperitoneal aerosol chemotherapy; FDG-PET/CT; Positron Emission Tomography scan; response evaluation
MeSH Terms: conditions — Peritoneal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: scan — Fluorodeoxyglucose (FDG)-positron emission tomography/Computed tomography scan

SUMMARY:
The pilot study will investigate the use of repeated FDG-PET/CT scans in 16 patients with peritoneal metastasis originating from abdominal cancers treated with Pressurized Intraperitoneal Aerosol Chemotherapy. The study will focus on the potential of repeated FDG-PET/CT scans to evaluate the treatment as well as the feasibility in the patient group.

DETAILED DESCRIPTION:
Background: Peritoneal metastasis (PM) is a late-stage manifestation of several gastro-intestinal cancers. Conventional administrated chemotherapy has limited effect due to the peritoneal-plasma barrier and most patients will die from their disease within a few months. An alternative treatment strategy, Pressurized IntraPeritoneal Aerosol Chemotherapy (PIPAC), has gained interest in the last decade. Prospective phase II studies have demonstrated significant local treatment effect and promising survival data initially within the palliative setting but more recently also with curative intent. The technical aspects of PIPAC are nearly uniform worldwide but there is no consensus on the optimal evaluation of treatment response. Currently, histological features in repeated biopsies from the peritoneum are used as an indicator of treatment response. Thus, easily accessible, and non-invasive alternatives are needed to optimize and personalize patient selection and to improve the response assessment. Both are also essential regarding future development and implementation of this treatment for both curative and palliative purposes. This could be achieved with the use of imaging techniques. Computed tomography (CT) scan holds well-known limitations in the detection of PM. Alternatively, several studies have investigated the use of the Positron emission tomography and CT (PET/CT) scans in the diagnostic setting of PM. This method shows promising results concerning visualization and assessing PM lesions, but no studies have investigated the ability of PET/CT scans to detect changes in PM during PIPAC treatment. Enabling the use of PET/CT scans as an evaluation tool for PIPAC-directed therapy is an important and necessary step to expand the clinical application. Also, non-invasive evaluation methods and consensus of evaluation is of significant importance for the quality of future randomized controlled trials in this field of research. We want to conduct a prospective study to investigate if PET/CT scans can detect changes within PM lesions in patients treated with PIPAC directed therapy. Since the study is the first of its kind, we plan to start with a pilot study including only a few patients. We will use the results to generate important knowledge for subsequent larger randomized studies on and clinical optimization of PIPAC directed therapy in patients with PM.

Objective: To investigate whether FDG-PET/CT scans can detect changes in PM in patients treated with PIPAC and whether the repeated scans are feasible within this group of patients.

Method: The pilot study will include 16 patients with known PM, four from each of the groups: gastric cancer, pancreatic cancer, colo-rectal cancer and ovarian cancer will be included. The patient will be offered standard PIPAC directed treatment (including standard histological evaluation of biopsies of the peritoneum) according to local guidelines. During the first series (one series is equivalent to three PIPAC treatments each five weeks) patients will receive three FDG-PET/CT's, one before PIPAC 1, one after PIPAC 2 and one after PIPAC 3. The scans will be described according to PERCIST (PET response criteria in solid tumors). In case of FDG-negative PM-disease at the first scan the patient will receive only one follow-up scan after PIPAC 2 to investigate whether the treatment if self can cause FDG-uptake in the PM elements.

ELIGIBILITY:
Inclusion Criteria:

* Patients with synchronous or metachronous histology or cytology proven GC, PC, CRC, or OC with clinical evidence of PM.
* Patients who are eligible for and offered PIPAC at the discretion of the dedicated multidisciplinary tumor conference and subsequent out-patient evaluation at Odense PIPAC Center
* Patients with a maximum of one extra-peritoneal metastasis at CT dated within one month of inclusion.
* Patients in Eastern Cooperative Oncology Group performance status 0-1.
* Patients >18 years of age.
* Patients must be able to give mandatory oral and written consent in Danish.

Exclusion Criteria:

* Concomitant systemic chemotherapy (bidirectional treatment).
* Known allergies to contrast dye.
* Any other significant disease or disorder which, in the opinion of the investigator, may either put the patient at risk because of participation in the trial, or may influence the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 16 patients with peritoneal metastasis, four from each of the groups: gastric cancer, pancreatic cancer, colo-rectal cancer and ovarien cancer, eligebel for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of patients with metabolic response according to FDG-PET/CT evaluated by PERCIST 1.0 one lesion after PIPAC 3 | 18 months
  The number of patients with metabolic response according to FDG-PET/CT evaluated by PERCIST 1.0 one lesion after PIPAC 3

SECONDARY OUTCOMES:
The number of patients with metabolic response after PIPAC 1 according to FDG-PET/CT evaluated by PERCIST 1.0 | 18 months
  The number of patients with metabolic response after PIPAC 1 according to FDG-PET/CT evaluated by PERCIST 1.0
The number of patients with changed treatment strategy due to extraperitoneal FDG-PET/CT findings after PIPAC 1 or PIPAC 3 | 18 months
  The number of patients with changed treatment strategy due to extraperitoneal FDG-PET/CT findings after PIPAC 1 or PIPAC 3
The number and reasons for discontinued FDG-PET/CT scans (feasibility) | 18 months
  The number and reasons for discontinued FDG-PET/CT scans (feasibility)
Number of patients with FDG-PET/CT positive peritoneal surface after PIPAC 1 despite negative baseline FDG-PET/CT (false positive/feasibility) | 18 months
  Number of patients with FDG-PET/CT positive peritoneal surface after PIPAC 1 despite negative baseline FDG-PET/CT (false positive/feasibility)
The number of patients where FDG-PET/CT evaluated by PERCIST one lesion agrees with histological response according to PRGS after PIPAC 1 and 3 | 18 months
  The number of patients where FDG-PET/CT evaluated by PERCIST one lesion agrees with histological response according to PRGS after PIPAC 1 and 3

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Mortensen, Professor, Study Director — Odense PIPAC Center, Department of Surgery, Odense University Hospital
Locations (1):
- Odense PIPAC Center, Odense, Funen, Denmark

IPD SHARING:
Plan to Share IPD: No
Publications and presentations will be based on patient data, but the database is not open to other researchers.